CLINICAL TRIAL: NCT02073695
Title: Return of Function and External Rotation Post Proximal Humerus Fracture Fixation With Neutral Rotation Brace
Acronym: ROTATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A publication released shortly after start indicating intervention not always beneficial. Fewer surgical cased thereafter.
Sponsor: Torbay and South Devon NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13/01/049
Record Dates: First submitted 2014-02-21; First posted 2014-02-27 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Proximal Humeral Fracture
Keywords: Proximal humeral fracture; Shoulder; Orthopaedics; Neutral rotation brace; Polysling
MeSH Terms: conditions — Shoulder Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neutral Rotation Brace (Other): Neutral Rotation Brace
  Interventions: Procedure: Operative procedure to fix proximal humeral; Device: Neutral Rotation Brace; Other: Physiotherapy review; Other: Functional outcome forms filled in; Other: Postal functional outcome scores; Other: Post-operative Radiographs
- Standard polysling (Current practice) (Other): Standard polysling (Current practice)
  Interventions: Procedure: Operative procedure to fix proximal humeral; Device: Neutral Rotation Brace; Other: Physiotherapy review; Other: Functional outcome forms filled in; Other: Postal functional outcome scores; Other: Post-operative Radiographs

INTERVENTIONS:
Procedure: Operative procedure to fix proximal humeral — Operative fixation by the shoulder team at Torbay Hospital
Device: Neutral Rotation Brace — Performed at the end of the surgical procedure at Torbay Hospital
Other: Physiotherapy review — Physiotherapy review on day of surgery, and post-surgery at 6 weeks, 3 months and 1 year.
Other: Functional outcome forms filled in
  Other Names: Oxford; DASH; SF-12
Other: Postal functional outcome scores — Sent to patient at 9 weeks post surgery
Other: Post-operative Radiographs — Performed at 6 weeks and 3 months at shoulder clinic appointment at Torbay Hospital

SUMMARY:
Research question:

Do patients using a neutral rotation brace post surgery have improved functional outcome and external rotation of the shoulder compared to current best practice using a polysling holding the proximal humerus in internal rotation?

Primary objectives:

To compare post-operative functional outcome scores obtained at 6 weeks, 9 weeks, 3 months and 1 year. (Scores at 6 weeks and 3 months in clinical review and postal scores at 9 weeks and 1 year) between patients held in neutral versus current standard rotation. These will be compared to scores taken pre-operatively.

Benefits:

There may be no extra benefits to patients from this trial however the results from the trial will help improve treatment for future patients at this hospital, and others across the country.

Risks/disadvantages:

The operation is the same in both groups studied, the study is investigating the use of the two different slings. The post-operative treatment is also the same, and all patients on the trial will receive the same amount of physiotherapy. It isn't anticipated that there will be any additional risk from this trial.

ELIGIBILITY:
Inclusion Criteria:

* Proximal humeral fractures requiring operative intervention with extramedullary plate fixation (i.e. fractures displaced by 1cm and/or angulated by 45 degrees or more)
* Age over 18 years of age
* Patient able to give informed consent

Exclusion Criteria:

* Patients having intra-operative findings to complete Pectoralis major rupture or if operative exposure requires complete Pectoralis major tenotomy. (These patients need to be held in internal rotation with a standard polysling to allow healing of the Pectoralis major tendon)
* Patients under 18 years of age
* Patients unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Oxford score | 1 Year post surgery
  Patients subjective assessment of pain and Activities of Daily Living (ADL) impairment. The Oxford Shoulder Questionnaire has been shown to correlate well with both the Constant Score and the SF36 assessment and to be sensitive to surgical intervention. The Oxford Shoulder Questionnaire accumulates to a total score with a maximum of value of 60, in which four pain related questions make up 33% of this total whilst the remaining 67% is derived from eight ADL related questions. The highest scores are attributed to the worst outcomes in the Oxford Shoulder Questionnaire
DASH - the Disabilities of the Arm, Shoulder and Hand | 1 year post surgery
  DASH Scoring system was developed to assess the level of disability for any patient with any condition affecting the upper limb by covering domains including symptoms, physical function and psychological function

SECONDARY OUTCOMES:
Range of movement(flexion, extension, abduction, external and internal rotation) | 6 weeks, 3 months and 1 year
  Assessed by Physiotherapists. Measurement will be performed using a goniometer to accurately assess range of movement
SF-12 Score | 1 Year post surgery
  This survey form has been shown to yield summary physical and mental health outcome scores
Range of movement (flexion, extension, abduction and internal rotation) | 6 weeks, 6 months and 1 year
  Conducted by physiotherapists. Measured using a goniometer to accurately assess range of movement
Time to union of fracture | 6 weeks and 3 Months
  X-Rays taken
Return to work post surgery | 1 year follow up
Re-operations and Complications | Throughout 1st year as applicable at outpatient appointments
  Documented at various outpatient appointments

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Conboy, FRCS (Orth), Principal Investigator — South Devon Healthcare
Locations (1):
- Torbay District General Hospital, Torquay, United Kingdom

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196